CLINICAL TRIAL: NCT03039335
Title: The Impact of Delayed Diagnosis of Alpha-1 Antitrypsin Deficiency: Assessing the Association Between Diagnostic Delay and Worsened Clinical Status
Brief Title: The Impact of Delayed Diagnosis of Alpha-1 Antitrypsin Deficiency
Status: Completed | Type: Observational
Sponsor: Biocerna LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 16001; Pro00019289 (Other: Chesapeake IRB)
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2018-07-16 (Actual); Status verified 2018-01

CONDITIONS: Alpha 1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with an AAT Deficiency: Subjects over the age of 18 that have been recently diagnosed with an Alpha-1 Antitrypsin deficiency will be enrolled into the study to observe the interval between first symptom and initial diagnosis.

SUMMARY:
The objective of this study is to prospectively assess whether there is any interval between first symptom and initial diagnosis that is experienced by patients with newly diagnosed alpha-1 antitrypsin deficiency (AATD) and then to assess whether this diagnostic interval is associated with worsened clinical status at the time of initial diagnosis.

DETAILED DESCRIPTION:
The study protocol proposes to assess participants' clinical status based on the results of spirometry tests that are performed by the patient's managing physician as a routine part of clinical care of individuals with AATD within +/- 6 months of the initial diagnosis, subjects' St. George's Respiratory Questionnaire (SGRQ) at the time of initial diagnosis, and their COPD Assessment Test (CAT) result at the time of initial diagnosis of AATD (hereafter called "time zero" or T0 defined as the day on which the patient's test shows AATD from the blood work submitted for testing to Biocerna LLC by the patients' managing physicians as part of their routine clinical management). After offering verbal consent, subjects will complete a survey that assesses various clinical domains, including demographic features, how was AATD ascertained, initial symptom ascribable to AATD, the number of healthcare providers (and specific types of providers) seen before initial diagnosis, and clinical status at T0 or within a defined, relatively narrow temporal window (+/- 6 months) of T0. As in prior studies, the diagnostic interval will be defined as the duration between self-reported initial symptom of AATD (usually dyspnea in > 80% of cases3) and initial confirmed diagnosis of AATD (T0).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Positive AATD Test Result

Exclusion Criteria:

* Previous Positive AATD Test Result
* Negative Test Result for AATD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AATD Positive Adult Subjects
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-04-15 (Actual)

PRIMARY OUTCOMES:
Recruitment | 3 months
  Track the number of subjects enrolled to determine if recruitment strategies need to be altered.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sanders, Principal Investigator — CEO of Biocerna LLC
Locations (1):
- Biocerna LLC, Fulton, Maryland, United States

IPD SHARING:
Plan to Share IPD: No